CLINICAL TRIAL: NCT06208514
Title: Brief Pain Exposure Therapy (BPET) For Nociplastic Pain
Acronym: BPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Sturgeon, Assistant Professor of Anesthesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00238637
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia; Lupus Erythematosus, Systemic; Chronic Pelvic Pain; Chronic Low Back Pain (CLBP)
Keywords: Pain exposure therapy; Telehealth-based behavioral intervention
MeSH Terms: conditions — Fibromyalgia; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: The enrollment numbers were increased to 125 (from 70) after the University of Michigan Medical School Institutional Review Board approved the amendment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief pain exposure therapy (BPET) (Experimental)
  Interventions: Behavioral: Brief pain exposure therapy (BPET)

INTERVENTIONS:
Behavioral: Brief pain exposure therapy (BPET) — Participants will complete daily logs for 7-days pre-treatment baseline, along with 21 days during the intervention protocol (fibromyalgia participants only will complete the daily logs), and 7 for days post-treatment.
  Brief Pain Exposure Therapy will be given for 3 weeks, 1.5 hours per week, telehealth-based behavioral intervention for chronic pain. Session content will include pain neuroscience education, mindfulness meditation, and graded exposure techniques for improving tolerance of painful or feared activities. Participants will also be provided handouts and pre-recorded meditation and imagery scripts that participants can use to facilitate between-session practices. In addition, participants will complete surveys through-out the study.

SUMMARY:
This study is intended to test whether a brief Zoom-based behavioral treatment can help adults with fibromyalgia (FM), Lupus, chronic pelvic pain, and chronic low back pain learn effective strategies for reducing pain, disability and other problems that can come with fibromyalgia, Lupus, chronic pelvic pain, and chronic low back pain (such as depression or anxiety).

DETAILED DESCRIPTION:
This project was amended and approved by the University of Michigan Medical School Institutional Review Board. These changes include adding chronic pelvic pain and chronic low back pain participants on to the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write and speak English
* Internet access and audio-visual conferencing capability (e.g., Zoom meetings by phone or computer) in the home

Fibromyalgia participants must have:

* Physician diagnosis of fibromyalgia
* OR: meet 2016 American College of Rheumatology (ACR) Criteria for FM: Widespread pain index score is ≥ 7 and symptom severity scale score is ≥ 5, or widespread pain index score is 4 to 6 and symptom severity score is ≥ 9
* OR: have pain self-reported in 4 out of 7 body regions in the General Sensory Sensitivity (GSS)-brief body map AND Opioid Use Disorder diagnosis by a physician.

Lupus participants must have:

* Physician diagnosis of systemic lupus erythematosus
* AND: Have pain self-reported in 4 out of 7 body regions in the GSS-brief body map
* AND: No change in medications or steroid dose for one month prior to entry (to avoid oscillation of steroid dosing during the study due to active disease).

Chronic Low Back Pain participants must have:

* Low Back Pain for at least half the days over the past 6 months
* Over the past 7 days, an average pain intensity of at least 4 out of 10

Exclusion Criteria:

* Indication of a co-occurring (non-fibromyalgia OR non-lupus) cause of chronic pain (e.g., inflammatory arthritis, other autoimmune disorders, spinal cord injury, cancer)
* Currently receiving cognitive-behavioral therapy or other psychological therapies for pain
* Open litigation regarding chronic pain in the past 1 year, as assessed in preliminary study screening.
* Inability to provide informed consent and complete study procedures (e.g., indications of suspected major cognitive impairment via observations of study staff during consenting) that would preclude comprehension or participation in study protocols.
* Pregnant or breastfeeding
* Any other diseases or conditions that would make a patient unsuitable for study participation as determined by the site principal investigators.
* Lupus group only: taking >10 mg prednisone (or equivalent steroid) dose per day as an indicator of ongoing disease activity (with no other strict exclusions based on medications)
* Chronic Pelvic Pain group only: surgery for any chronic pelvic pain related condition in the past 6 months
* Chronic low back pain only: scheduled back surgery; leg pain that is greater than your back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity based on the Numeric Pain Rating Scale between day 1 (T1) and day 60 (T5) | Day 1, Day 60
  This is a one item scale that participants answer worst pain experienced from no pain (0) to worst pain imaginable (10).

SECONDARY OUTCOMES:
Change in the Tampa Scale of Kinesiophobia (TSK) day 1 (T1) to day 60 (T5) | Day 1, Day 60
  This is a 17-item survey that participants answer strongly disagree (1) to strongly agree (4).
  Total scores are between 17-68 with a higher value indicating higher kinesiophobia.
Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference day 1 (T1) to day 60 (T5) | Day 1, Day 60
  Four questions are included in the PROMIS for pain interference. Participants will answer from not at all (1) to very much (5). Scores range from 4-20 with a higher score indicating more interference.
Change in pain intensity based on the Numeric Pain Rating Scale from day 1 (T1) to day 210 (T8) | Day 1, Day 210
  This is a one item scale that participants answer worst pain experienced from no pain (0) to worst pain imaginable (10).
Change in TSK from day 1 (T1) to day 210 (T8) | Day 1, Day 210
  This is a 17-item survey that participants answer strongly disagree (1) to strongly agree (4).
  Total scores are between 17-68 with a higher value indicating higher kinesiophobia.
Change in PROMIS Pain Interference from day 1 (T1) to day 210 (T8) | Day 1, Day 210
  Four questions are included in the PROMIS for pain interference. Participants will answer from not at all (1) to very much (5). Scores range from 4-20 with a higher score indicating more interference.
Acceptability of intervention based on Mean scores on the Treatment Acceptability and Adherence Scale (TAAS) | Day 29
  This is a 10-item survey that participant will complete after final intervention. Questions are answered from strongly disagree (1), neither agree or disagree (4), to agree (7). Scores above the midpoint - 35 out of 70 - will denote moderate acceptability of the intervention).
Feasibility based on the number of sessions attended | Day 29
  Higher number of sessions attended shows higher level of feasibility.
Feasibility based on the number of in-session and between-session practices completed | Day 29
  Higher number of sessions and between-sessions completed shows higher level of feasibility.
Feasibility based on open-ended feedback at the completion of the intervention | Day 29
  Participants will complete the open-ended feedback form that has 4 questions regarding the intervention and will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: John Sturgeon, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No